CLINICAL TRIAL: NCT07035652
Title: The Phase Ib Clinical Trial of the XH-S004 Tablet in Patients With Chronic Obstructive Pulmonary Disease (COPD) to Evaluate Its Safety, Tolerability, Pharmacokinetic Characteristics and Pharmacodynamic Characteristics After Multiple Administrations
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: S-INFINITY Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-S004-102
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Active neutrophil elastase
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1: Participant Group (Experimental): Up-titration design: prticipants received XH-S004 20 mg once daily (QD) from day 1 to day 28 in treatment period 1, XH-S004 40 mg once daily (QD) from day 29 to day 112 in treatment period 2, and XH-S004 60 mg once daily (QD) from day 113 to day 140 in treatment period 3.
  Pharmaceutical form: Tablets Route of administration: Oral
  Interventions: Other: XH-S004 20 mg, 40 mg or 60 mg
- Participant Group (Placebo Comparator): Participants received the matching placebo once daily (QD) from day 1 to day 140 in treatment period 1, treatment period 2 and treatment period 3.
  Pharmaceutical form: Tablets Route of administration: Oral
  Interventions: Other: Placebo

INTERVENTIONS:
Other: XH-S004 20 mg, 40 mg or 60 mg — Administered once per day for 140 days.
  Arms: Arm1: Participant Group
Other: Placebo — Administered once per day for 140 days.
  Arms: Participant Group

SUMMARY:
The objectives of the proposed study are to investigate safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and prliminary efficacy of XH-S004 in moderate to severe COPD patients with a stale standards of care (SOC).

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, placebo-controlled, up-titration study conducted in china, aimed at evaluating the safety and tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary efficacy of XH-S004 administered once daily for 140 days in COPD patients.

This study plans to enroll 81 COPD patients. Patients who sign the informed consent form will be screened according to the enrollment criteria, and randomly divided into 2 groups in 2:1 ratio (XH-S004 group: 54 participants and placebo group: 27 participants). Participants in XH-S004 group will receive XH-S004 20 mg for 28 days in treatment period 1, then up-titrated to XH-S004 40 mg for 84 days in treatment period 2, finally continue with XH-S004 60 mg for 28 days in treamtment period 3. Participants in placebo group will receive matching placebo from day 1 to day 140 (140 days in total).

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form (ICF);
2. Male or Female participants ages 40-80 (inclusive);
3. BMI ≥ 18.5 kg/m2 and ≤ 26 kg/m2, with male weight ≥50 kg and female weight ≥45 kg (inclusive);
4. Patients diagnosed with COPD according to 2024 GOLD consensus had a medical record or relevant documentation proving a history of COPD for ≥12 months at screening visit;
5. Current or former smokers with a smoking history of ≥10 pack-years;
6. Post-bronchodilator FEV1/ forced vital capacity [FVC] ratio <0.70 and post-bronchodilator FEV1 % predicted >30% and ≤70%.
7. Sputum volume≥10ml/day at screening visit;
8. with a documented history: 1) Moderate-to-severe COPD patients with a stable SOC therapy prior to signing ICF, including LABA, LAMA, LABA/LAMA, LABA/LAMA/ICS (evaluated by investigator to confirm the treatment regimen complies with clinical practice); Continuous use with a stable dosage for ≥1 month prior to randomization; Medication compliance between 80% and 120% from signing ICF to randomization; 2) Acute exacerbation history of ≥2 moderate or ≥1 severe requiring hospitalization within 12 months prior to screening.
9. Medical Research Council (MRC) Dyspnea Scale grade ≥2.
10. COPD Assessment Test (CAT)≥10

Exclusion Criteria:

1. Have a primary diagnosis of asthma as determined by the investigator;
2. During screening period, WBC<the lower limit of normal range, or absolute neutrophil count<the lower limit of normal range;
3. During screening period, blood eosinophils ≥300 cells/microliter;
4. Pregnant and lactating females

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-11-13 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced at Least One of Treatment-Related Adverse Events (AEs) or Serious Adverse Events (SAEs) | From randomisation to study completion, up to 168 days

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (Tmax) | From randomisation to study completion, up to 168 days
Maximum measured concentration (Cmax) of XH-S004 | From randomisation to study completion, up to 168 days
Maximum measured concentration of XH-S004 at steady state (Cmax,ss) | From randomisation to study completion, up to 168 days
Area Under the Plasma Concentration-time Curve (AUC) of XH-S004 | From randomisation to study completion, up to 168 days
Change From Baseline in Blood Concentration of Active Neutrophil Elastase (NE) | From randomisation to study completion, up to 168 days
Change from baseline in pre-brondilator FEV1 after first drug administration. | At baseline, day 28, day 112 and day 140
  FEV1 was used to assess lung function and is the maximum amount of air that can be forced out in one second after taking a deep breath.
Change from baseline in post-brondilator FEV1 after first drug administration | At baseline, day 28, day 112 and day 140
  FEV1 was used to assess lung function and is the maximum amount of air that can be forced out in one second after taking a deep breath.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No